CLINICAL TRIAL: NCT03746834
Title: NASHA/Dx as a Perianal Implant for the Treatment of Persistent Fecal Incontience After Anorectal Malformation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Johan Danielson, Principal investigator, Uppsala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 461:2013/6500
Record Dates: First submitted 2018-05-02; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Fecal Incontinence; Anorectal Malformation
Keywords: Fecal incontinence; Anorectal malformation
MeSH Terms: conditions — Fecal Incontinence; Anorectal Malformations

STUDY DESIGN:
Intervention Model Description: Patients are treated with injection of NASHA/Dx and act as their own Controls over time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Patients are given NASHA/Dx as a perianal injection
  Interventions: Device: NASHA/Dx (Solesta®)

INTERVENTIONS:
Device: NASHA/Dx (Solesta®) — Perianal submucosal injection of 3-4 ml of NASHA/Dx

SUMMARY:
Persistent fecal incontinence (FI) after anorectal malformations (ARM) is a common occurence. During the last two decades perianal injection therapy has emerged as an option for treating patients with FI due to other causes than ARMs. The studies done on different implants have always expempted patients with ARM which has led to ARM being a formal contraindication for treatment with perianal injection therapy.

The study aims to treat patients with persistent FI after ARM with perianal injection of NASHA/Dx (Solesta®) and follow them with Clinical examination and questionnaires up to 18 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Persistent FI (Miller incontinence score >5)
* Anorectal malformation.

Exclusion Criteria:

* Pregnancy
* Rectal prolapse
* Significant mucosal prolapse
* Inflammatory bowel disease
* Anorectal surgery within the last year Before inclusion
* Anticoagulant medication/bleeding diathesis
* Anorectal sepsis in the past
* Immunodeficiency
* Immunosuppressing therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2015-12-12 (Actual); Study Completion 2015-12-12 (Actual)

PRIMARY OUTCOMES:
Change in number of incontinence episodes | The change in number of incontinence episodes before treatment is compared with data at 18 months after injection.
  The number of incontinences episodes as measured over a two week interval The number of incontience episodes is measured with a bowel-movement-diary over a two week period.

SECONDARY OUTCOMES:
Miller´s incontinence score | Before treatment compared with data at 18 months after treatment. Miller´s incontinence score is measured on a scale from 0 (meaning total fecal continence) to 18 (meaning total fecal incontinence).
  Change of Miller´s incontinence score
Quality of life, general | Before treatment compared with data at 18 months after treatment. SF-36 measures quality of life in 8 subscales. Each scaled from 0 to 100. Higher score is considered better. Two total scores of mental and physical QoL can be calculated.
  Change in quality of Life as observed with SF-36
Adverse events | Before treatment compared with data at 18 months after treatment
  Control of any adverse events during the course of the study
Quality of life, disease specific | Before treatment compared with data at 18 months after treatment. Measures 4 subscales, each measuring 1-4. Higher score implies better quality of life.
  Change in quality of Life as observed with FIQL

IPD SHARING:
Plan to Share IPD: No
The data collected is of very personal type and since the number of subjects is so small there would be a risk of identification if all the data was released.

REFERENCES:
- [Result] Danielson J, Karlbom U, Wester T, Graf W. Efficacy and quality of life 2 years after treatment for faecal incontinence with injectable bulking agents. Tech Coloproctol. 2013 Aug;17(4):389-95. doi: 10.1007/s10151-012-0949-8. Epub 2012 Dec 7. PMID 23224913
- [Result] Danielson J, Karlbom U, Sonesson AC, Wester T, Graf W. Submucosal injection of stabilized nonanimal hyaluronic acid with dextranomer: a new treatment option for fecal incontinence. Dis Colon Rectum. 2009 Jun;52(6):1101-6. doi: 10.1007/DCR.0b013e31819f5cbf. PMID 19581853
- [Result] Danielson J, Karlbom U, Graf W, Wester T. Outcome in adults with anorectal malformations in relation to modern classification - Which patients do we need to follow beyond childhood? J Pediatr Surg. 2017 Mar;52(3):463-468. doi: 10.1016/j.jpedsurg.2016.10.051. Epub 2016 Nov 15. PMID 27894765